CLINICAL TRIAL: NCT04768868
Title: A Phase 1, Open-Label, Multi-Center, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of the WEE1 Inhibitor IMP7068 Monotherapy in Patients With Advanced Solid Tumors
Brief Title: The Safety and Pharmacokinetics Preliminary Efficacy of IMP7068 in Patients With Advanced Solid Tumors
Acronym: WEE1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Impact Therapeutics, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IMP7068 - 101
Record Dates: First submitted 2020-11-02; First posted 2021-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumors
Keywords: Breast Cancer; Ovarian Cancer; Prostate Cancer; Pancreatic Cancers
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Intervention Model Description: The dose schedules will be explored in this study (described below):
  Dose Schedule: IMP7068 administered QD on Days 1-3, Days 8-10 and Days 15-17 on a 21-day cycle.
  The other Dose Schedules may be explored according to SMC decision.
  The dose-expansion stage will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage. Approximately100 patients each with advanced solid tumor who has exhausted available treatment options with respective biomarker(s) determined by central laboratory will be evaluated. Single dosing will not be performed in the dose-expansion stage of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- IMP7068 (Other): Part 1: Dose Escalation
  The study will begin with open-label dose escalation in IMP7068 monotherapy treatment to determine the Maximum tolerated dose (MTD)
  Part 2: Dose Expansion The dose-expansion stage will commence after the Recommended Phase 2 Dose (RP2D) is determined during the dose-escalation stage. A total of 100 patients each with advanced solid tumor who has exhausted available treatment options will be evaluated.
  Interventions: Drug: IMP7068

INTERVENTIONS:
Drug: IMP7068 — To evaluate the safety tolerability, pharmacokinetics, and anti-tumor activity of the WEE1 inhibitor IMP7068 monotherapy in patients with advanced solid tumors

SUMMARY:
A Phase 1 Dose Escalation and Expansion Study of IMP7068 Monotherapy in Advanced Solid Tumors

DETAILED DESCRIPTION:
This is A Phase 1, Open-Label, Multi-Center, Dose Escalation and Expansion Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of the WEE1 Inhibitor IMP7068 Monotherapy in Patients with Advanced Solid Tumors

The study will include a dose-escalation stage and a dose-expansion stage. The dose-escalation stage is designed to determine the maximum tolerated dose (MTD) and select recommended Phase 2 dose (RP2D) of IMP7068 monotherapy. The dose-expansion stage will be conducted with RP2D to further evaluate the preliminary anti-tumor activity, safety and tolerability.

A total of approximately 140-350 patients will be enrolled in the study.

Approximately 60-100 patients will be enrolled into Part 1 dose escalation of IMP7068 monotherapy. A total of 100 patients each with advanced solid tumor will be evaluated in Part 2 dose-expansion of IMP7068 monotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. The patient must voluntarily participate in this clinical study. Be willing and able to provide written informed consent form (ICF) prior to any study activity.
2. Age ≥18 years on the day of signing the ICF, males or females. Only for Korea, Age ≥19 years on the day of signing the ICF.
3. The enrolled patients must have histologically or cytologically confirmed advanced solid tumor that is refractory/intolerant to standard treatment or for which no standard treatment exists. The patients with known microsatellite-instability high (MSI-H) or deficient in mismatch repair (dMMR) disease are required to have received prior PD 1/PD-L1 therapy; those with known NTRK fusion are required to have received an approved TRK-inhibitor. The patients who are suitable for resection or other localized therapy that is potentially curative are not eligible.

Key Exclusion Criteria:

1. Patients with active or untreated known CNS metastases and/or carcinomatous meningitis should be excluded.
2. Patients with serious acute or chronic infections.
3. Patients who have received prescription or non-prescription drugs or other products known to be sensitive to CYP3A4 substrates or CYP3A4 substrates with a narrow therapeutic index, or to be moderate to strong inhibitors/inducers of CYP3A4 which cannot be discontinued 7 days prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of IMP7068.
4. Patients who are participating in or have participated in a study of an investigational agent and received study therapy or used an investigational device within 28 days of the first dose of treatment.
5. Patients have not recovered (i.e., to Grade ≤1 or to baseline, as evaluated by NCI-CTCAE Version 5.0) from prior anti-cancer therapy-induced AEs, except for alopecia, anorexia or CTCAE grade 2 peripheral neuropathy.
6. Patients who have undergone a major surgery or have undergone a radical radiotherapy within 28 days prior to the study treatment, or have undergone a palliative radiotherapy within 14 days prior to the study treatment, or have used a radioactive drug (Strontium, Samarium, etc.) within 56 days prior to the study treatment.
7. Patients who are unable to swallow oral medications. Patients have gastrointestinal illnesses that may clinically significantly affect the absorption of oral medication IMP7068 at discretion of investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-02-25 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Part 1 Dose Escalation: Incidence of treatment emergent adverse events (TEAEs) | Day 1 through to 30 days after last dose (approximately 4 cycles (84 days plus 30 day follow-up )); Each cycle is 21 days
Part 1 Dose Escalation: Severity of treatment emergent adverse events (TEAEs), according to the National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE), version 5.0 | Day 1 through to 30 days after last dose (approximately 4 cycles (84 days plus 30 day follow-up )); Each cycle is 21 days
Part 1 Dose Escalation: Recommended Phase 2 Dose (RP2D) of IMP7068 monotherapy | Day 1 through to start of dose expansion phase (approximately 1 year)
  Recommended Phase 2 Dose (RP2D) of IMP7068 monotherapy (selected by the safety monitoring committee (SMC) based on pharmacokinetics, target saturation at steady state, pharmacodynamics, safety, tolerability and preliminary anti-tumor effects of the dose range studied)
Part 2 Dose Expansion: Overall Response Rate (ORR) | Day 1 through 30 days after last dose, estimated to be 5 months
  Overall Response Rate (ORR) for all cohorts (percentage of patients who had a best response rating of complete response (CR) and partial response (PR), according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, which was maintained ≥4 weeks)

SECONDARY OUTCOMES:
Plasma Concentration of IMP7068 | Day -7 to repeat dose Day 1; postdose at multiple time points from Day 1 to Day 21 in Cycle 1 (Cycle 1 = 21 days), Day 1 on Cycle 2 (Cycle 2 onwards = 21 day-cycles) and subsequent cycles (Up to 26 months)
Part 1 Dose Escalation: Objective response rate (ORR): percentage of patients who had a best response | Within the first year: every 6 weeks, thereafter every 12 weeks to end of treatment (EOT) visit (approximately 84 days), documented disease progression, withdrawal of consent, loss to follow-up, death or termination of the study (whichever occurs first)
Part 1 Dose Escalation: Progression-free survival (PFS): duration of time from date of first dose to date of disease progression (according to RECIST v1.1) or death due to any cause, whichever comes first) | Within the first year: every 6 weeks (±7 days); thereafter: every 12 weeks (±7 days); or when clinically indicated (Approximately 1 year )
Part 1 Dose Escalation: Overall survival (OS): time from date of first dose to death due to any cause | Every 12 weeks±14 days after the last dose, until up to 2 years, withdrawal of consent, loss to follow-up, death, or termination of the study, whichever occurs first
Part 1 Dose Escalation: Duration of response (DOR): duration of time a patient is evaluated as either complete response (CR) or partial response (PR) as best response until the first date that the criteria for progression are met, or death. | Day 1 through 30 days after last dose, estimated to be 5 months
Part 1 Dose Escalation: Disease control rate (DCR): proportion of patients who had a best response rating of complete response (CR) or partial response (PR), or stable disease (SD), which was maintained ≥6 weeks from Day 1 of Cycle 1 | Day 1 through 30 days after last dose, estimated to be 5 months
Part 2 Dose Expansion: Progression-free survival (PFS) duration of time from date of first dose to date of disease progression (according to RECIST v1.1) or death due to any cause, whichever comes first) | Day 1 through 30 days after last dose, estimated to be 5 months
Part 2 Dose Expansion: Duration of response (DOR) duration of time a patient is evaluated as either CR or PR as best response until the first date that the criteria for progression are met, or death | Day 1 through 30 days after last dose, estimated to be 5 months
Part 2 Dose Expansion: Incidence of Treatment emergent adverse events (TEAE) | Day 1 through 30 days after last dose, estimated to be 5 months
Part 2 Dose Expansion: Severity of Treatment emergent adverse events (TEAE) according to the NCI-CTCAE, version 5.0 | Day 1 through 30 days after last dose, estimated to be 5 months

CONTACTS AND LOCATIONS:
Locations (16):
- United States (7):
  - Emory University Hospital, Atlanta, Georgia
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Mary Crowley Cancer Research, Dallas, Texas
  - Next Oncology, San Antonio, Texas
- China (4):
  - Wuhan Union Hospital, Wuhan, HB
  - West China 2nd University Hospital, Chengdu, Sichuan
  - Beijing Cancer Hospital, Beijing
  - Fudan University Shanghai Cancer Center, Shanghai
- Taiwan (5):
  - Chang Gung Medical Foundation - Linkou Branch, Taoyuan District, TW
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Hospital, Liouying, Tainan
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No